CLINICAL TRIAL: NCT01515670
Title: Length of Stay and Complications in High-risk Patients Receiving Fast-track Total Hip (THA) or Knee- Alloplasty (TKA).
Status: Completed | Type: Observational
Sponsor: Rigshospitalet, Denmark (Other)
Collaborators: Hvidovre University Hospital (Other); Aarhus University Hospital (Other); Vejle Hospital (Other); Esbjerg Hospital - University Hospital of Southern Denmark (Other); Regional Hospital Holstebro (Other); Naestved Hospital (Other); Bispebjerg Hospital (Other); Central Jutland Regional Hospital (Other); Aalborg University Hospital (Other)
Responsible Party: Principal Investigator, Christoffer Joergensen, Research-fellow, Rigshospitalet, Denmark
Other Study IDs: RH30-0623
Record Dates: First submitted 2012-01-18; First posted 2012-01-24 (Estimated); Last update posted 2021-06-22 (Actual); Status verified 2021-06

CONDITIONS: Arthroplasty Complications; Co-morbidity; Postoperative Morbidity
Keywords: THA; TKA; Fast-track; Enhanced recovery; preoperative co-morbidity; postoperative morbidity; Arthroplasty; Replacement; Hip; Knee; Morbidity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 90 Days
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Fast-track THA/TKA: Any patient receiving THA/TKA in the participating wards

SUMMARY:
The purpose of the study is to determine the influence of preoperative co-morbidity in relation to increased length of stay and postoperative complications in patients receiving fast-track hip or knee replacement.

DETAILED DESCRIPTION:
Preoperative risk assessment is well established and repeatedly demonstrated to be related to adverse postoperative outcomes regarding all organ functions. However, all evidence is based upon conventional care programs and none has been done on fast-track surgery, neither in total hip arthroplasty (THA) or total knee arthroplasty (TKA).

The purpose of this study series is therefore to evaluate the importance of conventional risk factors in an optimised fast-track TKA and THA set-up. These studies will be performed in the Lundbeck Foundation Center for fast-track THA and TKA, based on an established database, but with additional detailed risk information to be included in studies of certain types co-morbidity.

The Lundbeck Foundation Center Database prospectively registers patient characteristics and co-morbidity in all patients receiving hip and knee arthroplasty. This is done using a questionaire and with dedicated staff available to help in case of doubt regarding specific questions. Additional information is collected by scrutinizing the patients medical charts. Completeness of data has been shown to be about 95%.

ELIGIBILITY:
Inclusion Criteria:

* Standardized elective fast-track THA or TKA

Exclusion Criteria:

* Elective THA or TKA not in regular fast-track setup
* not a Danish citizen

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: unselected patients receiving THA or TKA
Sampling Method: Probability Sample
Enrollment: 60000 (Actual)
Dates: Start 2010-02 (Actual); Primary Completion 2019-01 (Actual); Study Completion 2019-01 (Actual)

PRIMARY OUTCOMES:
Length of hospital stay and reasons for length of hospital stay >4days | At discharge
  Number of nights spend in hospital after day of surgery, including transferral between departments.
  Any procedure followed by more than 4 days in hospital will have review of discharge papers to determine causes of the "prolonged" admission
Surgically related readmissions | 90 days after surgery
  Evaluation of any potentially surgery related readmission 90 days after discharge. Readmissions defined as related are defined as: Revision due to prosthesis problems, deep venous thrombosis (DVT), pulmonary embolism (PE) (verified or disproved), stroke/transitory cerebral ischaemia (TCI), possible wound infection (return to operating theatre, treatment with antibiotics only, no treatment), fractures without known trauma, falls, knee manipulation, hip dislocation, cardiac problems (acute myocardial infarction (AMI), any type of arrhythmia), pneumonia, urinary retention (UR), abdominal complications (gastric ulcer, ileus) and sequelae (rehabilitation, opioid side-effects, pain, other conditions related to surgery). Readmissions due to chronic obstructive lung disease (COPD), syncope and urinary tract infection (UTI) ≤ 30 days of primary admission

SECONDARY OUTCOMES:
Mortality 90 days after surgery | 90 days after surgery
  Evaluation of all deaths 90 days after surgery

OTHER OUTCOMES:
Co-morbidity related readmissions | 90 days after surgery
  Depending on the type of co-morbidity investigated, special attention and analysis of readmissions found to be related to the specific type of co-morbidity will be done

CONTACTS AND LOCATIONS:
Overall Officials: Christoffer C Joergensen, MD, Principal Investigator — Rigshospitalet, Denmark
Locations (7):
- Denmark (7):
  - Himmerland Hospital, Farsø, Judland
  - Holstebro Regionalhospital, Holstebro, Judland
  - Vejle Hospital, Vejle, Judland
  - Hvidovre Hospital, Hvidovre, Region Sjælland
  - Bispebjerg University Hospital, Copenhagen
  - Gentofte University Hospital, Gentofte Municipality
  - Næstved Hospital, Næstved

REFERENCES:
- [Derived] Ortved M, Petersen PB, Jorgensen CC, Kehlet H; Lundbeck Foundation Centre for Fast-track Hip and Knee Replacement Collaborative Group. Postoperative Morbidity and Mortality in Diabetic Patients After Fast-Track Hip and Knee Arthroplasty: A Prospective Follow-up Cohort of 36,762 Procedures. Anesth Analg. 2021 Jul 1;133(1):115-122. doi: 10.1213/ANE.0000000000005248. PMID 33234944
- [Derived] Jorgensen CC, Gromov K, Petersen PB, Kehlet H; Lundbeck Foundation Centre for Fast-track Hip and Knee Replacement Collaborative Group. Influence of day of surgery and prediction of LOS > 2 days after fast-track hip and knee replacement. Acta Orthop. 2021 Apr;92(2):170-175. doi: 10.1080/17453674.2020.1844946. Epub 2020 Nov 12. PMID 33176546
- [Derived] Petersen PB, Jorgensen CC, Kehlet H; Lundbeck Foundation Center for Fast-track Hip and Knee Replacement collaborative group. Temporal trends in length of stay and readmissions after fast-track hip and knee arthroplasty. Dan Med J. 2019 Jul;66(7):A5553. PMID 31256778
- [Derived] Jorgensen CC, Petersen MA, Kehlet H; Lundbeck Foundation Centre for Fast-Track Hip and Knee Replacement Collaborative Group. Preoperative prediction of potentially preventable morbidity after fast-track hip and knee arthroplasty: a detailed descriptive cohort study. BMJ Open. 2016 Jan 12;6(1):e009813. doi: 10.1136/bmjopen-2015-009813. PMID 26758264